CLINICAL TRIAL: NCT06974448
Title: Comparison of Frontal Hemodynamic Responses and Electrical Brain Activity During Dual Tasks in COPD Patients Versus Healthy Individuals
Brief Title: Hemodynamic Responses and Brain Activity During Dual Tasks in COPD Patients Versus Healthy Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melike Meşe Buran, MSc, PT, Hacettepe University
Other Study IDs: SBA 24/860
Record Dates: First submitted 2025-01-03; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease; Healty Controls
Keywords: COPD - Chronic Obstructive Pulmonary Disease; dual task; cognitive function; electroencephalogram; Functional Near-Infrared Spectroscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COPD Group
- Control Group

SUMMARY:
Abstract

Cognitive dysfunction is joint in patients with chronic obstructive pulmonary disease (COPD).

In particular, there are effects in tasks that require attention, executive functions, and working memory related to the prefrontal cortex. These effects make it difficult to perform two tasks simultaneously and cause performance errors. The number of studies investigating the effects of cognitive impairments on dual-task performance in COPD is limited. In these studies, no tests were applied specifically for attention and working memory areas; therefore, the brain's neural activity was not investigated during these tests. Multimodal approaches are recommended for a comprehensive assessment of the functional activity of the brain. Multimodal approaches provide more accurate results than single-modality approaches. In the integrated electroencephalography (EEG)-functional near-infrared spectroscopy (fNIRS) approach, EEG provides adequate temporal resolution, while fNIRS offers better spatial resolution and is robust to noise. There is no study in COPD where simultaneous fNIRS-EEG measurements were made during both cognitive tests and dual tasks. In our study, the simultaneous measurement of frontal hemodynamic responses and electrical brain activity in both cognitive tests and dual-task conditions and the examination of the relationship between the results and arterial stiffness, balance, exercise capacity, anxiety, depression, and quality of life scores, which are reported to be related to cognitive function in COPD, constitute the original aspect of our study. The study will include 16 COPD and 16 healthy individuals. The same assessments will be made in both groups, and the results will be compared. General and task-specific cognitive tests, prefrontal cortex oxygenation (fNIRS), electrical brain activity (EEG), exercise capacity, muscle oxygenation, arterial stiffness, balance, respiratory function, dyspnea, depression, anxiety, and quality of life will be evaluated. As a result of this study is expected to determine the effects of cognitive function and dual-task on frontal hemodynamic responses and electrical brain activity in COPD.

DETAILED DESCRIPTION:
This study aims to compare frontal hemodynamic responses and electrical brain activity to a dual task in individuals with COPD and healthy individuals and to investigate the relationship between frontal hemodynamic response and electrical brain activity and exercise capacity, arterial stiffness, balance, depression, anxiety, or quality of life.

The required sample size for the project was calculated as 28 individuals, 14 each for the COPD and control groups (G*Power Version 3.1.9.4, Franz Faul, Universitat Kiel, Germany), with a statistical significance of 94% test power and 0.05 error level for a difference of 3.33 points and 2.59 standard deviation (effect size 1.455) in the Mini-Mental State Examination score assessing cognitive function between the COPD and control groups. Considering a 10% dropout rate for each group, a total of 32 individuals, 16 in each group, will be included in the study.

Exercise tests will be performed with at least one day of rest breaks.

1. st Session

   * Patient file information will be recorded.
   * A respiratory function test will be performed.
   * MoCA and MMDT tests will be performed to evaluate general cognitive status.
   * 6DWT tests will be performed. Muscle oxygenation will be measured during the test.
   * An SGRQ questionnaire will be administered to the COPD Group.
   * NHP questionnaire will be performed.
2. nd Session

   * Arterial stiffness measurement will be performed.
   * TUG test will be performed.
   * The HAD scale will be applied
   * Cardiopulmonary exercise capacity will be evaluated. Muscle oxygenation will be measured during the test.
3. rd Session

   * Task-specific cognitive tests, Stroop tests, and N-back tests will be performed. fNIRS and EEG measurements will be performed during the Stroop and N-back tests.
   * fNIRS and EEG measurements will be made during single and dual tasks.

Data Collection: The researchers will collect data on frontal hemodynamic responses, electrical brain activity, exercise capacity, arterial stiffness, and balance parameters through tests. Data on dyspnea, depression, anxiety, and quality of life measurements will be collected through scales applied during face-to-face interviews.

Data Analysis: Statistical analysis of the data obtained from all volunteers included in the study will be performed using the IBM SPSS 24.0 (SPSS Inc, Chicago, USA) program. Descriptive statistics will be calculated. The conformity of the variables to normal distribution will be evaluated using visual (histogram and probability graphs) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). In comparisons between groups, Student t-test will be used when parametric test assumptions are met, and Mann Whitney U test will be used when parametric test assumptions are not met. Chi-square test will be used for comparisons of categorical variables. Correlation between data that are normally distributed will be analyzed using Pearson correlation, and those that are not normally distributed will be analyzed using Spearman correlation. The error probability will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria for the COPD Group:

* Being diagnosed with COPD
* Being between the ages of 40-65
* Not having a history of exacerbations in the last 4 week
* Being willing to participate in the study

Inclusion criteria for the Control Group

* Being between the ages of 40-65
* Being willing to participate in the study

Exclusion Criteria for COPD Group :

* Known alpha-1 anti-trypsin deficiency
* Presence of ischemic heart disease, uncontrolled hypertension, and diabetes mellitus
* Presence of obstructive sleep apnea syndrome
* Untreated tumors
* Known history of dementia
* Existing musculoskeletal, neuromuscular, or neurological diseases that may prevent participation in the tests
* Not being willing to participate in the study

Exclusion criteria for the Control Group:

* Having a known chronic health problem
* Not being willing to participate in the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who were followed up at Hacettepe University Chest Diseases Department due to COPD diagnosis and referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit for physiotherapy and rehabilitation (COPD Group).
  Individuals with COPD (COPD Group) and healthy individuals who were matched in terms of age and gender and volunteered to participate in the study (relatives of the researchers, relatives of the patients, and hospital staff) (Control Group).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMST) | through study completion, an average of 1 year
  The Mini-Mental State Examination (MMST) will be used for general cognitive status assessment.
  MMST consists of 11 items grouped under five main headings (execution, recording memory, attention and calculation, recall and language). The total score is obtained by adding the scores obtained by the patient from each item. It is evaluated out of a total of 30 points.The Turkish version of the test will be used
Montreal Cognitive Assessment Scale (MoCA) | through study completion, an average of 1 year
  MoCA, the presence of cognitive impairment will be evaluated using the MoCA scale. The scale is scored between 0 and 30 points. The application time of the scale is approximately 10 minutes and includes six cognitive functions. The cognitive functions evaluated in the scale are memory, visual-spatial skills, executive functions, attention, concentration and working memory tasks, language and orientation. The Turkish version of the scale will be used.
Stroop test | through study completion, an average of 1 year
  The Stroop test is a widely used test to evaluate executive functions of the frontal region, such as selective attention, information processing speed, cognitive flexibility, and the ability to resist interference. It is one of the tests considered the gold standard for measuring a person's attention. It is especially preferred to measure executive control in a situation that creates cognitive conflict. In the Stroop test, the person is expected to shift their attention to the color of the ink the word is written in, rather than the semantic meaning. When there is a conflict between visual information (the color of the ink the word is written in) and semantic information (the meaning of the word), the person's response is delayed or gives an incorrect answer.
N back test | through study completion, an average of 1 year
  The N-back test has been used in both experimental and neuroimaging studies as a measure of working memory ability and has been called the gold standard technique for the assessment of working memory. The study will use a "0-back and 2-back task". During this test, the participant is expected to respond if the stimulus shown on the screen overlaps with the stimulus shown 'n' times before. Various letters were selected as stimuli. The visual stimulus appeared on the screen for 500 milliseconds (msec), with a 2000 msec waiting period between the two stimuli. All participants will be initially informed about the task, then given a practice test, and will proceed to the main test after at least three correct responses. No intervention will be made during the main test. In the evaluation of this test, the number of correct hits and false alarms will be determined according to the participant's responses, and correct hit and false alarm scores will be calculated using these data.
Evaluation of hemodynamic responses in brain oxygenation | through study completion, an average of 1 year
  Functional Near Infrared Spectroscopy (fNIRS) will evaluate hemodynamic responses in brain oxygenation. FNIRS examinations measure hemodynamic responses (oxyhemoglobin and deoxyhemoglobin) in brain oxygenation to be able to transmit physical activity. It is a non-invasive optical imaging technique that allows real-time assessment of brain capacity. This will be an economical, high-durability (Artinis, Brite, Netherlands) wired 27-channel dual-wave length (760 and 850 nm) continuous wave (CW-fNIRS) system. Measurement will be performed during the cognitive , single and dual tasks.
Evaluation of Changes in Brain Electrical Activity-Electroencephalography (EEG) | through study completion, an average of 1 year
  EEG is a measurement of electrical activity in the brain that records the frequencies observed during normal brain activity. EEG signals will be collected using a 32-channel EEG device (Mobile EEG Enobio, Neuroelectrics, Barcelona, Spain), portable, wireless data acquisition system at a sample rate of 250 Hz. The EEG device will be synchronized using e-PRIME (Physiology Software Tools. Brain waves are divided into delta (0-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), low beta (12-16 Hz), high beta (16-25 Hz) and gamma (25-50 Hz) waves.The constituent factors of cognitive load will be measured separately in terms of the degree of activation of brain waves according to frequency. Measurement will be performed during the cognitive, single and dual tasks.

SECONDARY OUTCOMES:
Demographic Assessment | baseline
  The participants' age, gender, height, body weight, and smoking will be recorded. Clinical data will be recorded from the patients' file information, including COPD diagnosis period, risk factors, and COPD stage. The participants' accompanying diseases will be evaluated with the Charlson Comorbidity Index, developed to predict chronic diseases' effect on mortality and morbidity.
Charlson Comorbidity Index | baseline
  Charlson Comorbidity Index is calculated by giving coronary artery disease, congestive heart failure, peripheral vascular diseases, cerebrovascular diseases, dementia, chronic lung disease, connective tissue disease, peptic ulcer disease, mild liver disease, diabetes "1 point", hemiplegia, moderate or severe kidney disease, diabetes causing end-organ damage, any tumor presence, leukemia, lymphoma "2 points", moderate or severe liver disease "3 points", metastatic solid tumor, AIDS "6 points". As the comorbidity score increases, the risk of mortality and morbidity increases in patients.
Forced expiratory volume in one second | through study completion, an average of 1 year
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Forced vital capacity | through study completion, an average of 1 year
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Forced expiratory volume in one second/forced vital capacity ratio | through study completion, an average of 1 year
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/forced vital capacity ratio will be recorded.
Forced mid-expiratory flow (FEF25-75) | through study completion, an average of 1 year
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded.
Peak expiratory flow | through study completion, an average of 1 year
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Evaluation of Dyspnea | through study completion, an average of 1 year
  Dyspnea will be evaluated with the Modified Medical Research Council dyspnea scale (MMRC). The MMRC evaluates patients' shortness of breath during a specific situation such as walking, climbing a hill or stairs. The scale is read aloud to patients and they are asked to mark the most appropriate option. The MMRC is a categorical scale used to describe individuals' dyspnea levels, with five statements ranging from 0 to 4 points, where the most appropriate statement regarding shortness of breath is selected. Higher scores indicate greater dyspnea severity.
Functional Capacity Assessment | through study completion, an average of 1 year
  The 6-Minute Walk Test (6MWT) will be performed to assess functional capacity. For the 6MWT, individuals are asked to walk in a 30-meter corridor at the maximum speed they can walk without running. The test will be repeated twice at a 30-minute interval, and the distance covered at the end of the second test will be recorded in meters.
Assessment of Maximal Exercise Capacity | through study completion, an average of 1 year
  Maximal exercise capacity will be determined by cardiopulmonary exercise testing (CPET). The protocol will be performed on a bicycle ergometer (Lode Corival, Groningen, Netherlands) in accordance with the European Respiratory Society's criteria. Cardiopulmonary responses and effort perceptions will be recorded.
Evaluation of muscle oxygenation (SmO2) levels | through study completion, an average of 1 year
  During CPET and 6MWT, muscle oxygenation (SmO2) levels will also be measured. SmO2 level will be assessed with a wearable muscle oxygenation measurement device (Moxy, Fortiori Design LLC, Minnesota, USA) that measures local oxygen saturation in muscle capillaries. The device will be placed on the quadriceps muscle. The SmO2 level will be measured as a percentage, and the difference between the starting and ending percentages of the test will be recorded as a percentage.
Arterial Stiffness Assessment | through study completion, an average of 1 year
  Arterial stiffness will be assessed with a portable measuring device (Tel-O-Graph BT, IEMGmbh, Aachen, Germany). Measurement will be performed in a quiet room after 12 hours of fasting in the morning, in a sitting position, with the patient resting for 15 minutes. Measurements will be performed three times at five-minute intervals.
Functional Balance Assessment | through study completion, an average of 1 year
  The Timed Up Go Test (TUG) will be performed for functional balance assessment. In the TUG test, the participant is asked to get up from the chair without support, walk three meters, and then return to the chair without support. At the end of the test, the number of seconds it took the individual to complete the test will be recorded. The test will be performed twice, and the best score obtained from the two attempts will be recorded.
Assessment of Anxiety and Depression Levels | through study completion, an average of 1 year
  The Hospital Anxiety and Depression Scale (HAD) will be used to assess anxiety and depression levels. HAD scale has been used in many studies on COPD. The total score ranges from 0 to 21 points, with scores <14 considered "normal." The scale's validity and reliability study was conducted, and the Turkish population-adapted form will be used.
St. George's Respiratory Questionnaire (SGRQ) | through study completion, an average of 1 year
  St. George's Respiratory Questionnaire (SGRQ) will be used to assess disease-specific quality of life. The "symptoms" section (29 items) includes items related to symptom level, sputum production, cough frequency, breathlessness, wheezing or frequency and duration of wheezing attacks. The "Activity" section (9 items) evaluates physical activities that are restricted due to shortness of breath or that cause shortness of breath. The final section, the "Impact" section (38 items), evaluates factors such as panic, health checks, medication requirements and side effects, work, daily life effects and expectations for health. Each section is scored separately between 0-100 points. A "0 point" indicates that there is no impairment in quality of life.A validity and reliability study of the questionnaire was conducted, and an adapted form for the Turkish population will be used. The scale will be applied only to the COPD Group.
Nottingham Health Profile (NHP) | through study completion, an average of 1 year
  The Nottingham Health Profile (NHP) will assess general quality of life. The NHP is a general quality of life scale developed to measure perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire, which consists of a total of 38 items, evaluates six different parameters related to health status. These parameters are physical activity (8 items), emotional reactions (9 items), energy (3 items), social isolation (5 items), pain (8 items) and sleep (5 items). Each subparameter is scored between 0-100. A higher score indicates a worsening health status.The scale's validity and reliability study was conducted, and the Turkish population's adapted form will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Mese- Buran, Msc, PT., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Polatli M, Yorgancioglu A, Aydemir O, Yilmaz Demirci N, Kirkil G, Atis Nayci S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Validity and reliability of Turkish version of St. George's respiratory questionnaire]. Tuberk Toraks. 2013;61(2):81-7. doi: 10.5578/tt.5404. Turkish. PMID 23875584
- [Background] Zhang L, Sun J, Sun B, Luo Q, Gong H. Studying hemispheric lateralization during a Stroop task through near-infrared spectroscopy-based connectivity. J Biomed Opt. 2014 May;19(5):57012. doi: 10.1117/1.JBO.19.5.057012. PMID 24862561
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Kaygusuz MH, Oral Tapan O, Tapan U, Genc S. Balance impairment and cognitive dysfunction in patients with chronic obstructive pulmonary disease under 65 years. Clin Respir J. 2022 Mar;16(3):200-207. doi: 10.1111/crj.13469. Epub 2022 Jan 26. PMID 35081270
- [Background] Alvarez-Bueno C, Cunha PG, Martinez-Vizcaino V, Pozuelo-Carrascosa DP, Visier-Alfonso ME, Jimenez-Lopez E, Cavero-Redondo I. Arterial Stiffness and Cognition Among Adults: A Systematic Review and Meta-Analysis of Observational and Longitudinal Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014621. doi: 10.1161/JAHA.119.014621. Epub 2020 Feb 28. PMID 32106748
- [Background] Li R, Yang D, Fang F, Hong KS, Reiss AL, Zhang Y. Concurrent fNIRS and EEG for Brain Function Investigation: A Systematic, Methodology-Focused Review. Sensors (Basel). 2022 Aug 5;22(15):5865. doi: 10.3390/s22155865. PMID 35957421
- [Background] Reijnders T, Troosters T, Janssens W, Gosselink R, Langer D, Davenport PW, von Leupoldt A. Brain Activations to Dyspnea in Patients With COPD. Front Physiol. 2020 Jan 24;11:7. doi: 10.3389/fphys.2020.00007. eCollection 2020. PMID 32038311
- [Background] Hassan SA, Bonetti LV, Kasawara KT, Beal DS, Rozenberg D, Reid WD. Decreased automaticity contributes to dual task decrements in older compared to younger adults. Eur J Appl Physiol. 2022 Apr;122(4):965-974. doi: 10.1007/s00421-022-04891-w. Epub 2022 Jan 27. PMID 35084541
- [Background] Hassan SA, Campos MA, Kasawara KT, Bonetti LV, Patterson KK, Beal DS, Fregonezi GAF, Stanbrook MB, Reid WD. Changes in Oxyhemoglobin Concentration in the Prefrontal Cortex during Cognitive-Motor Dual Tasks in People with Chronic Obstructive Pulmonary Disease. COPD. 2020 Jun;17(3):289-296. doi: 10.1080/15412555.2020.1767561. Epub 2020 May 22. PMID 32441147
- [Background] Gore S, Blackwood J, Ziccardi T. Associations Between Cognitive Function, Balance, and Gait Speed in Community-Dwelling Older Adults with COPD. J Geriatr Phys Ther. 2023 Jan-Mar 01;46(1):46-52. doi: 10.1519/JPT.0000000000000323. Epub 2021 Jul 29. PMID 34334706
- [Background] Wen XH, Li Y, Han D, Sun L, Ren PX, Ren D. The relationship between cognitive function and arterial partial pressure O2 in patients with COPD: A meta-analysis. Medicine (Baltimore). 2018 Jan;97(4):e9599. doi: 10.1097/MD.0000000000009599. PMID 29369175
- [Background] Higbee DH, Dodd JW. Cognitive impairment in COPD: an often overlooked co-morbidity. Expert Rev Respir Med. 2021 Jan;15(1):9-11. doi: 10.1080/17476348.2020.1811090. Epub 2020 Aug 26. No abstract available. PMID 32811226
- See also: GLOBAL STRATEGY FOR PREVENTION, DIAGNOSIS AND MANAGEMENT OF COPD: 2023 Report — https://goldcopd.org/2023-gold-report-2/